CLINICAL TRIAL: NCT01345435
Title: A Multi-center, Randomized, Parallel, Interventional, Open Label Trial to Compare Hemoglobin A1C-lowering Effect of Conventional Treatment and Smart Care Service in Patients With Type 2 Diabetes
Brief Title: Effects of Telemonitoring and Telemedicine Service for Type 2 Diabetes Care
Acronym: Smart-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHANGHEE LEE (Industry)
Collaborators: LG Electronics Inc. (Industry); Purdue University (Other)
Responsible Party: Sponsor-Investigator, CHANGHEE LEE, Chief Research Engineer, LG Electronics Inc.
Organization: LG Electronics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Smartcare-DM
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes
Keywords: telemonitoring; usual care; telemedicine; telehealth; home care; Health Care Quality; Access; Evaluation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Telemonitoring group (Experimental): * A Smart Care PC, blood glucose meter and body composition analyzer will be provided
  * transmitting the results to the Smart Care Server via Smart Care PC
  * At Smart care Center,care manager will provide remote blood glucose monitoring and individual diabetes case management
  Interventions: Procedure: Telemonitoring group
- Telemonitoring & Telemedicine group (Experimental): * A Smart Care PC, blood glucose meter and body composition analyzer will be provided
  * transmitting the results to the Smart Care Server via Smart Care PC
  * At Smart care Center,care manager will provide remote blood glucose monitoring and individual diabetes case management
  * taking telemedicine through video telephone instead of visiting hospital
  Interventions: Procedure: Telemonitoring & Telemedicine
- Control group (Other): * Blood glucose meter and body composition analyzer will be provided
  * Self-monitoring Blood Glucose (SMBG)
  Interventions: Other: SMBG

INTERVENTIONS:
Procedure: Telemonitoring group — The Telemonitoring group will be provided blood glucose meter, body composition analyzer, and remote monitoring PC. They should visit the site once per every 2 months (8 weeks), and measure their blood glucose using a provided blood glucose monitor twice a day during study period (once after first morning urination and once before going to bed). After measurement of blood glucose and body composition, the subjects should make transmit measured information through Smart Care PC into a centralized server of Smart Care Center. At Smart care Center, care manager will provide remote blood glucose monitoring and individual diabetes case management
  Other Names: Smartcare System : Telemonitoring
  Arms: Telemonitoring group
Procedure: Telemonitoring & Telemedicine — The Telemonitoring & Telemedicine group will be provided blood glucose meter, body composition analyzer, and remote monitoring PC. They should measure their blood glucose using a provided blood glucose monitor twice a day during the study period. After measurement of blood glucose and body composition, the subjects should make transmit measured information through Smart Care PC into a centralized server of Smart Care Center. At Smart care Center, care manager will provide remote blood glucose monitoring and individual diabetes case management. A remote medical doctor should provide medical consultation to the subjects through videotelephony using the remote monitoring PC and then issue electronic prescriptions.
  Other Names: Smartcare System : Telemonitoring & Telemedicine
  Arms: Telemonitoring & Telemedicine group
Other: SMBG — The subjects who are assigned in the control group will be provided blood glucose Monitor. The subjects who are assigned in the control group should perform the same blood glucose measurement same as the test group during the study, and measured results should be recorded in a diary of self blood glucose measurement. In addition, the subjects should visit the site once per every two months (8 weeks).
  Other Names: Self blood glucose measurement
  Arms: Control group

SUMMARY:
A multi-center, randomized, parallel, interventional, open label trial to compare Hemoglobin A1C-lowering effect of conventional treatment and Smart Care Service in patients with type 2 diabetes.

DETAILED DESCRIPTION:
1. Objectives : To evaluate superiority in the Hemoglobin A1C -lowering effect of Smart Care Service compared to the conventional treatment in patients with type 2 diabetes.
2. Test and control group

   * Control group : The subject group who is receiving any conventional treatment (hospital visit).
   * Test groups

     * Conventional treatment + remote monitoring group: The subject group who is receiving the health care services using conventional treatment (hospital visit) and remote monitoring.
     * Remote visit + remote monitoring group: The subject group who is receiving remote visit and remote monitoring using videotelephony
3. Target Subject: Type II diabetes patients

ELIGIBILITY:
Inclusion Criteria:

1. More than 20 years of age and under 60 years of age
2. Patients who are able to receive outpatient treatment with type II diabetes mellitus.
3. If the patients require using insulin, patients who are using basal insulin or premixed insulin less than 2 times a day are eligible.
4. Patients with HbA1c above 7% and less than 11% (7%≤HbA1c≤11%).
5. Patients who are able to understand the purpose of this trial and to read and write.
6. Patients who are able to use the Smart Care PC for this study.
7. Patients who have wired/wireless internet access at home.
8. Patients who participate voluntarily and sign the informed consent.

Exclusion Criteria:

1. Patients with type I diabetes mellitus
2. Patients who are using Bolus insulin (short-acting insulin) or insulin pump.
3. Patients who take medicines which can significantly affect glycemic control.
4. Patients with acute illness, untreated other disease or diabetic complications required additional treatment.
5. Patients currently being hospitalized or planning to hospitalize during the study period.
6. Patients who have severe renal disease (above 1.5 times the upper limit of normal serum creatinine levels).
7. Pregnant or lactating women.
8. Patients with any severe liver disease including cirrhosis (AST or ALT: above 3 times the upper limit of normal).
9. Patients with uncontrolled chronic lung disease.
10. Patients with known history of alcoholism, mental illness, or drug dependency.
11. Patients who have cognitive disorder or psychiatric problems
12. Patients who have participated in other clinical trial within 12 weeks prior to screening visit.
13. Any clinically significant medical condition including neurologic disease, gastrointestinal disease or malignant tumor, etc., which may affect the test results, or any other medical condition which in the opinion of the investigator makes the patients unsuitable for participation in the trial.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 417 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in Hemoglobin A1c | 0 and 24 weeks
  Changes in Hemoglobin A1c from baseline to 24 weeks visit.
  Reduce Hemoglobin A1c after study

SECONDARY OUTCOMES:
Changes in FBS (Fasting blood sugar) | 0 and 24 weeks
  Changes in FBS (Fasting blood sugar) from baseline to 24 weeks visit
  Maintains FBS within the normal range
Changes in lipid profile | 0 and 24 weeks
  Changes in lipid profile from baseline to 24 weeks visit
  Maintains normal lipid profile
Percentage of subjects who achieved goal Hemoglobin A1c | 0 and 24 weeks
  Goal Hemoglobin A1c <7%
Changes in body mass index (BMI) | 0 and 24 weeks
  Reduction of body mass index
  - BMI=Body weight (kg)/Height2(m)
SMBG(Self-monitoring of blood glucose) compliance | up to 24 weeks
  measurement of Self-monitoring of blood glucose
Changes in body weight | 0 and 24 weeks
  Reduce body weight from baseline to 24 weeks visit
Assessment of patients' satisfaction | 24 weeks
  Assessment of subjects' satisfaction, Only remote monitoring group and remote visit + remote monitoring group are applicable
Medication compliance | up to 24 weeks
  * Patients diary will be recorded and medication compliance will be calculated by calculating the number of days administered Insulin or Oral Hypoglycemic Agents during the study
  * Drugs compliance = the number of days administered antihypertensive drugs / participated period in this study * 100%

CONTACTS AND LOCATIONS:
Overall Officials: In Kyu Lee, M.D., Principal Investigator — Kyungpook National University Hospital
Locations (4):
- South Korea (4):
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Gangnam Severance Hospital, Seoul
  - Yonsei University Health System, Seoul